CLINICAL TRIAL: NCT04348994
Title: 3-year Follow up of Patients With Stress Urinary Incontinence Treated With Minimally Invasive Er: YAG Laser
Brief Title: Long-term Effectiveness of Non-ablative Er: YAG Laser for Treatment of Stress Urinary Incontinence (SUI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adrian Gaspar (Other)
Collaborators: Fotona d.o.o. (Industry)
Responsible Party: Sponsor-Investigator, Adrian Gaspar, Principal Investigator, Espacio Gaspar Clinic
Organization: Espacio Gaspar Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUI/01/2015
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; non-ablative Er:YAG laser
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser therapy (Experimental): Non-ablative thermal-only Er:YAG laser treatment using IncontiLase® protocol.
  Interventions: Device: Non-ablative thermal-only Er:YAG laser therapy

INTERVENTIONS:
Device: Non-ablative thermal-only Er:YAG laser therapy — Each patient will receive 3 sessions of Er:YAG laser treatment for SUI (IncontiLase®).
  Single-session treatments will be offered to patients after 18, 24 and 30 months following the initial three sessions.
  Other Names: IncontiLase®

SUMMARY:
Study is designed to assess the long-term clinical effects and safety profile of non-ablative Er:YAG (IncontiLase®) laser treatment, the durability of the results and the optimal treatment regimen for mild-to-severe stages of genuine female stress urinary incontinence (SUI).

DETAILED DESCRIPTION:
All patients with urodynamically proven SUI, who have failed/declined conservative therapies will be informed about the study.

They will be invited to attend a screening/baseline visit. At this visit, they will be asked to perform a standardised 1 hour pad test. Their medical history will be checked and they will undergo a clinical and vaginal examination, pregnancy test and dip stick urinalysis. If their 1 hour pad weight is >2g and they meet all other inclusion / exclusion criteria, they will be eligible for inclusion. They will receive detailed instructions for performing a 24 hour pad test, and will be asked to keep a 3 day voiding diary. They will be given the International Consultation on Incontinence Questionnaire Short Form (ICIQ-UI SF).

Patients will then undergo 3 outpatient treatment visits. The timing of visits will be approximately 1 month apart. At each of their 3 outpatient appointments, they will be asked about any deleterious effects since their last appointment. Patients will receive 3 treatments in total.

Patients will be invited to attend a follow-up visits 3, 6, 12 and 18 months after the 3rd treatment and asked to complete the 1 hour pad test, 24 hour pad test, 3 day voiding diary and ICIQ-SF questionnaire.

At the 18-, 24- and 30-month follow up, they will be given an option to receive additional single session of non-ablative Er:YAG laser treatment. At each visit, and during additional visit after 36 months, they will be asked to complete all of the tests (1 hour pad test, 24 h hour pad test, 3 day voiding diary and ICIQ-UI SF).

ELIGIBILITY:
Inclusion Criteria:

* Adult Female, 18 years of age or older
* Clinical and urodynamic study (UDS) diagnosis of Stress Urinary Incontinence
* No significant improvement in urinary incontinence from at least one previous conservative treatment, such as pelvic floor muscle training

Exclusion Criteria:

* Pre-existing bladder pathology including prior radiation treatment
* Pregnancy
* BMI>35
* Radical pelvic surgery or previous incontinence surgery
* Urinary tract infection or other active infections of urinary tract or bladder
* SUI III (VLPP > 60 cm H2O)
* Any form of pelvic organ prolapse (POP) stage 2 or greater, according to POP-Q
* Diagnosis of urge incontinence
* Diagnosis of collagen disorders eg.benign joint hypermobility / Elhers-Danlos / Marfans etc.
* Incomplete bladder emptying
* Vesicovaginal fistula
* Faecal incontinence
* Unwillingness or inability to complete follow-up schedule
* Unwillingness or inability to give Informed Consent
* Failure to comply with diary requirements during extended baseline period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of ICIQ-UI SF scores | Baseline, 3, 6, 12, 18, 24, 30 and 36 months
  Change in mean test scores range = 0 - 21; low score = mild symptoms, high score = significant impact on quality of life.
Assessment of 1 hour pad weight test | Baseline, 3, 6, 12, 18, 24, 30 and 36 months
  The change in standardised 1 hour pad weight test from baseline to 36 months following treatment schedule.

SECONDARY OUTCOMES:
Change in 24 hour pad weight test | Baseline, 3, 6, 12, 18, 24, 30 and 36 months
  The change in standardised 24 hour pad weight test from baseline to 36 months following treatment schedule.
Change in leakage frequency as assessed by 3 day voiding diary | Baseline, 3, 6, 12, 18, 24, 30 and 36 months
  The change in leakage frequency from baseline to 36 months following treatment schedule.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaspar A, Koron N, Silva J, Brandi H. Vaginal erbium laser for treatment of stress urinary incontinence: optimization of treatment regimen for a sustained long-term effect. Lasers Med Sci. 2022 Jun;37(4):2157-2164. doi: 10.1007/s10103-021-03474-z. Epub 2022 Jan 24. PMID 35067817